CLINICAL TRIAL: NCT03502850
Title: A Phase I/II Study to Assess the Safety,Tolerability, Pharmacokinetics and Anti-tumour Activity of ASK120067 in Patients With Locally Advanced or Metastatic T790M Mutation-positive Non-Small Cell Lung Cancer Who Have Progressed Following Prior Therapy With an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Agent
Brief Title: Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of ASK120067 in Locally Advanced and Metastatic Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASK-LC-120067-Ⅰ/Ⅱ
Record Dates: First submitted 2018-04-10; First posted 2018-04-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASK120067 (Experimental): patients take ASK120067 orally once per day at different dose
  Interventions: Drug: ASK120067

INTERVENTIONS:
Drug: ASK120067 — patients take ASK120067 orally once per day at 40,80,160,240,320,480mg

SUMMARY:
ASK120067 Tablets is a Epidermal Growth Factor Receptor (EGFR) mutation selective Tyrosine Kinase Inhibitor which can efficient suppress the EGFR T790M drug-resistant mutation tumor cell in Xenograft mouse model. This study aims at local advanced or metastatic non-small cell lung cancer patients with T790M drug-resistant mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged from 18 years older to 70.
* Histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC
* Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including at least one of G719X, exon 19 deletion, L858R, L861Q mutation)
* Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI e.g. gefitinib or erlotinib or Afatinib, or Icotinib (Third EGFR TKI are not included). In addition other lines of therapy may have been given
* Documented evidence of definitely EGFR T790M+ state in the tumor tissue after disease progression on the most recent treatment regimen (irrespective of whether this is EGFR TKI or chemotherapy)
* At least one lesion, not previously irradiated and not chosen for fresh biopsy during the study screening period, that can be accurately measured at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short access ≥ 15mm) with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
* ECOG performance status of 0 to 2.
* Life expectancy of at least 12 weeks
* Females should not be in lactation period and must have a negative pregnancy test prior to start of dosing; During the whole treatment,all patients should be in the entire 3 months during and after the treatment, repeated barrier precautions.
* Male patients were to be willing to use barrier contraception, ie, condoms and avoid sperm donation within 6 months
* Signed consent on an Independent Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation

Exclusion Criteria:

* Any Target cancer drug from a previous treatment regimen or clinical study within 8 days, or less than approximately 5x half-life of the first dose of study treatment
* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs （including traditional Chinese medicine）from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment
* The third EGFR-TKI from a previous treatment regimen or clinical study (ie, AZD9291, CO-1686, HM61713, avitinib,BPI-15086,BPI-7711,Alflutinib,Almonertinib)
* Major surgery within 4 weeks of the first dose of study treatment
* Radiotherapy with a wide field of radiation or bone marrow radiotherapy is more than 30% within 4 weeks of the first dose of study treatment
* Taking (or cannot stop taking 1 week before the first dose receiving) strong inhibitor of CYP3A4
* With the exception of alopecia and grade 2 or higher, prior platinum-therapy related neuropathy, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 2 at the time of starting study treatment
* Spinal compression, or brain metastasis exhibiting symptoms but untreated (except those exhibit no symptom with stable condition and do not apply corticosteroids for 4 weeks before the trail initiating)
* Any evidence showing severe or inadequate controlled systemic disease. For example patients with inadequate controlled hypertension or active hemorrhagic tendency considered not suitable for the trail or would affect the compliance towards the protocol
* Active infection such as HBV (HBV-DNA≥1000cps/ml), HCV, HIV, syphilis et al .
* Any condition affecting the drug taking, or significantly affecting the absorption or the pharmacokinetic parameters, include any kind of uncontrollable nausea or vomit, chronic gastroenteropathy, disability in swallowing, and history of gastrointestinal resection or surgery
* Any condition meet the following cardiac standard: Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 ECG. All kinds of abnormal in cardiac rhythm, conduction and resting ECG profile with clinical significance, for example complete left bundle branch block, 2 or 3 grade of conduction block and a PR interval>250 msec. Any possible factors increasing the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval. left ventricular ejection fraction (LVEF) within 40%.
* Any history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonia require steroid therapy or active interstitial lung disease with clinical evidence during recruiting
* Hyperglycemia that cannot be stably controlled by drugs (fasting blood glucose is greater than or equal to 7.0mmol/L)
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: Absolute neutrophil count < 1.5 x 109/L. Platelet count < 100 x 109/L. Haemoglobin < 90 g/L. Alanine aminotransferase> 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases. Aspartate aminotransferase > 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases. Total bilirubin > 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN.
* History of hypersensitivity to active or inactive excipients of ASK120067 or drugs with a similar chemical structure or class to ASK120067
* Women who were breastfeeding and pregnant
* Any other cancer, within 5 years prior to screening with the exception of adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin, or papillary thyroid cancer
* Judgment by the investigator that any serious or uncontrolled eye disease may increase the safety risk of the patient .
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years.
  Evaluation of objective response rate assessed by RECIST 1.1

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events | Adverse events will be collected from baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, ophthalmic examinations and NCI CTCAE v4.03
Progression free survival | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival
Duration of response | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years.
  Duration of response assessed by RECIST 1.1
Disease control rate | CT or MRI at screening and every 2 Cycles (from first dose of multiple dosing) until disease progression,date of death or withdrawal from study,whichever came first, assessed up to approximately 2 years.
  Evaluation of Disease control rate assessed by RECIST 1.1
Overall survival | Time from treatment start to the time of death due to any cause or withdrawal from study,whichever came first, assessed up to approximately 2 years.
  defined as the time from date of first dose until date of death due to any cause
Maximum Plasma Concentration [Cmax] of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out Cmax
Peak Plasma Time [tmax] of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out tmax
Area under the plasma concentration versus time curve (AUC) of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day1 to figure out AUC
Terminal rate constant of single dose single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out terminal rate constant
Clearance of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out clearance
Half life of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out half life
Volume of distribution of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of f ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out volume of distribution
Mean resistance time of single dose ASK120067 | Blood samples will be collected from each subject at pre-specified times after the first dose of the study on Day 1, (pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24, 48, 72 ,96,144 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolite following single dose at designated time points of Day 1 to figure out mean resistance time
Steady state Cmax of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Cmax of ASK120067 and 1 metabolite at steady state following multiple doses
Steady state tmax of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Tmax of ASK120067 and 1 metabolite at steady state following multiple doses
Steady state Cmin (Minimum Plasma Concentration) of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Cmin of ASK120067 and 1 metabolite at steady state following multiple doses
Steady state AUC of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  AUC of ASK120067 and 1 metabolite at steady state following multiple doses
Steady state clearance of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Clearance of ASK120067 and 1 metabolite at steady state following multiple doses
Accumulation ratio of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Accumulation ratio of ASK120067 and 1 metabolite following multiple doses
Time dependency of multiple doses ASK120067 | Blood samples will be collected from each subject at pre-specified times during the multiple dosing cycles (Cycle 1-pre-dose Day 8, 10,12,15,18,22. Cycle 1 D28- pre-dose, 1, 2, 3, 4, 5,6, 8, 10, 24 hours post dose)
  Time dependency of ASK120067 and 1 metabolite following multiple doses

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Li B, Wu L, Pan Y, Pan Z, Liu Y, Fan Y, Ji Y, Fang J, Shi Q, Shi J, Gao H, Hu Y, Wang X, He Z, Ma R, Zhang Y, Jiang D, Bai Y, Zhang Y, Huang L, Zhou T, Liu H, Wang D, Wen Q, Chen G, Zang A, Wang X, Zhang X, Hu J, Yang R, Zhang G, Gu K, Wang L, Wang Q, Wei Z, Li Z, Lu H, Zhang H, Chen H, Song T. Efficacy and Safety of Limertinib (ASK120067) in Patients With Locally Advanced or Metastatic EGFR Thr790Met-Mutated NSCLC: A Multicenter, Single-Arm, Phase 2b Study. J Thorac Oncol. 2022 Oct;17(10):1205-1215. doi: 10.1016/j.jtho.2022.05.011. Epub 2022 Jun 2. PMID 35659581